CLINICAL TRIAL: NCT06432556
Title: Study of Cellular Heterogeneity in Patients With Mastocytosis (MastCellHet) Mastocytosis Cell Heterogeneity
Brief Title: Study of Cellular Heterogeneity in Patients With Mastocytosis
Acronym: MastCellHet
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/23/0362; 2024-A00021-46 (Other: ID-RCB)
Record Dates: First submitted 2024-04-29; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Mastocytosis
Keywords: Mastocytosis; Mast cells; Cellular heterogeneity; CD 45+; CD 34+
MeSH Terms: conditions — Mastocytosis | interventions — Single-Cell Gene Expression Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- patients with isolated cutaneous mastocytosis with associated skin involvement - RNAseq (Other)
  Interventions: Genetic: scRNAseq; Procedure: two Skin biopsies
- patients with mastocytosis indolent systemic with associated skin involvement (Other)
  Interventions: Procedure: one Skin biopsies
- patients with isolated cutaneous mastocytosis with associated skin involvement (Other)
  Interventions: Procedure: one Skin biopsies
- patients with mastocytosis indolent systemic with associated skin involvement - RNAseq (Other)
  Interventions: Genetic: scRNAseq; Procedure: two Skin biopsies

INTERVENTIONS:
Genetic: scRNAseq — A blood test tube (only for scRNAseq, 2 tubes of 10 ml per patient)
  Arms: patients with isolated cutaneous mastocytosis with associated skin involvement - RNAseq; patients with mastocytosis indolent systemic with associated skin involvement - RNAseq
Procedure: two Skin biopsies — 2 skin biopsies from a lesional area
  Arms: patients with isolated cutaneous mastocytosis with associated skin involvement - RNAseq; patients with mastocytosis indolent systemic with associated skin involvement - RNAseq
Procedure: one Skin biopsies — 1 skin biopsies from a lesional area
  Arms: patients with isolated cutaneous mastocytosis with associated skin involvement; patients with mastocytosis indolent systemic with associated skin involvement

SUMMARY:
This study will aim to study the heterogeneity of skin-resident mast cells and of blood circulating hematopoietic progenitors in patients suffering from isolated Cutaneous Mastocytosis and from systemic Mastocytosis with skin lesions.

DETAILED DESCRIPTION:
Mastocytosis is a rare disease caused by abnormal mast cell accumulation/proliferation. Its clinical features are very heterogeneous. Among adult patients, 15% present an isolated cutaneous mastocytosis (CM), while 85% of them present a systemic mastocytosis (SM) with cutaneous lesions. In addition, regardless of the diagnosis (i.e., CM or SM), it is frequent to observe mast cell-dependent symptoms of variable severity, ranging from gastrointestinal discomfort to life-threatening reactions. To date, the origin of such heterogeneous manifestations in adult patients is still elusive. Researchers hypothesize that the heterogeneity in mastocytosis symptoms might originate, at least in part, from a broad diversity of mast cell populations in patients. This study will aim to uncover heterogeneity of skin-resident mast cells and of blood circulating hematopoietic progenitors in patients suffering from isolated CM or SM with skin lesions. Patients with isolated CM and patients with SM with cutaneous involvement will be recruited from the Mastocytosis Expert Center of Toulouse.

Cluster of Differentiation (CD) 45+ cells from skin biopsies and CD 34+ cells from blood will be isolated by magnetic cell sorting for scRNAseq. Bioinformatics analysis pipeline will be used in order to analyze the cellular heterogeneity of skin lesions and blood from CM and SM patients by comparing their transcriptomic signatures. Using trajectories analysis, the researchers will then deduce infer a differentiation pathway between blood progenitors and cutaneous mast cells at the patient level. Researchers will then confirm the expression of identified relevant biomarkers by highly multiplexed imaging in frozen skin biopsies from CM patients and from SM patients.

ELIGIBILITY:
Inclusion Criteria:

* Criteria related to the study population:
* Subject affiliated with a social security or insurance scheme
* Subject who has given written consent to his participation in the study
* Criteria related to the studied pathology:
* Subject diagnosed with isolated cutaneous or indolent systemic mastocytosis with associated skin involvement defined according to World Health Organization criteria (and/or international criteria for cutaneous mastocytosis)
* Subjects whose KIT mutation status is known in the skin, bone marrow, and blood

Exclusion Criteria:

* Criteria related to the study population:
* Sun exposure of the biopsied areas expected within the 4 weeks preceding
* Subjects who have had exposure to sunlight or artificial UV radiation within the 2 weeks preceding inclusion at the biopsied areas
* Adult patients under legal protection, guardianship, or curatorship
* Pregnant or lactating women
* Criteria related to the studied pathology:
* Subjects with an advanced version of the pathology or advanced systemic mastocytosis (SAMA)
* Subjects with a known history of allergy or intolerance to local anesthetics
* Subjects who have previously shown abnormalities in skin healing or any other contraindication to skin biopsy
* Subjects with recognized addiction to alcoholism or drug abuse
* Subjects with a hereditary or acquired disorder of hemostasis
* Subjects with a severe or acute chronic condition judged by the investigator as incompatible with the trial
* Subjects presenting a clinically incompatible immune deficiency with the study
* Patients without a well-established diagnosis of mastocytosis
* Patients included in a therapeutic study for indolent systemic mastocytosis
* Treatment-related criteria:
* Any topical or systemic treatment for atopic dermatitis (including phototherapy) ongoing or stopped at least 14 days before the inclusion visit
* Systemic corticosteroids within the 4 weeks preceding the inclusion visit
* Ongoing systemic treatment likely to interfere with the healing process
* Subjects who have undergone physical treatment (radiotherapy, etc.) on the biopsy area in the past 6 months
* History of treatment or concomitant treatment that may interfere with the conduct of the study as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Study of the diversity of skin CD 45+ cells and circulating blood CD 34+ cells | 24 month and one week
  This study aims to examine the diversity of CD 45+ cells in the skin and CD 34+ cells in the circulating blood in patients. The approach used will be single cell sequencing (scRNAseq) to identify the transcriptomic profiles of the different cell populations in these two types of mastocytosis.

SECONDARY OUTCOMES:
Study of common or differential transcripts | 24 month and one week
  This part of the study will focus on analyzing common or differential genetic transcripts between patients with isolated cutaneous mastocytosis and those with systemic mastocytosis. The aim is to understand the underlying molecular differences between these two forms of the disease.

OTHER OUTCOMES:
marker | 24 month and one week
  through advanced imaging techniques (multiplexed imaging), marker in patients with isolated cutaneous mastocytosis and systemic mastocytosis will be identified compared with control sample
marker - isolated cutaneous mastocytosis | 24 month and one week
  through advanced imaging techniques (multiplexed imaging), marker in patients with isolated cutaneous mastocytosis will be identified compared with control sample
marker - systemic mastocytosis | 24 month and one week
  through advanced imaging techniques (multiplexed imaging), marker in patients with systemic mastocytosis will be identified compared with control sample

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Bulai Livideanu, MD, Principal Investigator — Toulouse univiversity hospital
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No